CLINICAL TRIAL: NCT01537380
Title: Tissue and Plasma Pharmacokinetics of Cefazolin in Antibiotic Prophylaxis in Bariatric Surgery, an Open Label, Prospective, Single Center Trial
Brief Title: Tissue and Plasma Pharmacokinetics of Cefazolin in Antibiotic Prophylaxis in Bariatric Surgery
Acronym: Cefasleeve
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BRD/11/06-R
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Bariatric Surgery
MeSH Terms: interventions — Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cefazoline (Experimental)
  Interventions: Drug: Cefazoline

INTERVENTIONS:
Drug: Cefazoline — Injection of CEFAZOLINE (4 grams) 30-60 min before skin incision. A second injection will performed every 4 hours during the surgery

SUMMARY:
With 6.5 million obese recorded in France in 2009, obesity is a major public health: it is a chronic disease associated with many respiratory, cardiac, metabolic, musculoskeletal complications. The risk of mortality and morbidity are directly proportional to the importance of overweight and medical treatment alone is only moderately effective weight loss. Bariatric surgery is the only treatment with proven efficacy in patients with a body mass index above 40 kg/m2. As with any surgery, there is a risk of surgical site infection (SSI). The SSI are the third most common nosocomial infection after urinary tract infections and airway. The fight against the ISO requires the administration of antibiotic prophylaxis acting on the main bacteria found in bariatric surgery. There are several studies in the literature interested in the dose of cefazolin in bariatric surgery. However, no published pharmacokinetic studies defines an optimal dose to obtain tissue and plasmatic concentrations of cefazolin higher than minimum inhibitory concentrations of the main germs encountered in these surgery. Only empirical recommendations are published, including the SFAR and the National Institute of Health in 2010. This study aims to determine whether the dose of 4 grams of cefazolin can achieve these goals of concentration and estimate an injection time of preoperative ideal for an adequate tissue concentration at the time of the incision.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged > 18 years.
* BMI ≥ 40 and ≤ 65 kg/m2.
* The patient has given informed consent in writing.

Exclusion Criteria:

* Age less than 18 years and above 70 years.
* Major Trust.
* Pregnancy.
* Moderate to severe renal insufficiency or clearance creatinine clearance <60 ml / min
* Hypersensitivity to cephalosporins and beta-lactams.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Tissue concentration of cefazolin in the superficial subcutaneous fat during the surgical procedure | At the time of incision (T0), 1 hour of operation (T1), and at the closure (T2)

SECONDARY OUTCOMES:
Cefazolin tissue concentrations in fatty deep peri gastric tissue throughout the intervention | At the time of incision (T0), 1 hour of operation (T1), and at the closure (T2)
Kinetics of tissue concentrations of the superficial subcutaneous fat during surgery in patients with BMI < 50 and patients with BMI > 50 | At the time of incision (T0), 1 hour of operation (T1), and at the closure (T2)
Kinetics of tissue concentrations of the deep fat peri gastric during surgery in patients with BMI < 50 and patients with BMI > 50 | At the time of incision (T0), 1 hour of operation (T1), and at the closure (T2)
Kinetics of plasma concentrations during surgery in each group | At the time of incision, at 15, 30, 60 minutes of operation, and at the closure
Number of SSI following the surgery. | Within 30 days post-surgery
Area Under Curve (AUC) of cefazolin plasma kinetics for each group | Surgical incision,15,30,60 minutes post-incision, surgical closure

CONTACTS AND LOCATIONS:
Overall Officials: Romain Dumont, MD, Principal Investigator — Nantes Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Cinotti R, Dumont R, Ronchi L, Roquilly A, Atthar V, Gregoire M, Planche L, Letessier E, Dailly E, Asehnoune K. Cefazolin tissue concentrations with a prophylactic dose administered before sleeve gastrectomy in obese patients: a single centre study in 116 patients. Br J Anaesth. 2018 Jun;120(6):1202-1208. doi: 10.1016/j.bja.2017.10.023. Epub 2017 Dec 6. PMID 29793587